CLINICAL TRIAL: NCT07129317
Title: Pediatric Radiation Therapy Registry
Status: Recruiting | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Clark Charitable Foundation Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: J2563; IRB00504065 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Sarcoma; Pediatric Brain Tumors
Keywords: Pediatric; Brain tumor; Registry; Proton radiation; Radiation therapy; Photon radiation
MeSH Terms: conditions — Sarcoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pediatric brain tumors: Pediatric patients diagnosed with brain tumors requiring treatment with either proton or photon radiation therapy.
- Pediatric sarcomas: Pediatric patients diagnosed with bone or soft tissue sarcomas requiring treatment with either proton or photon radiation therapy.
- Non-brain-tumor and non-sarcoma

SUMMARY:
The Johns Hopkins Pediatric Radiation Oncology Program is creating a registry that will capture the full 3D radiation dosimetry delivered to its pediatric patients to manage the quality of care provided, as well as to examine the long-term outcomes and toxicity of each patient. The registry will capture baseline clinical data, disease, toxicity, and quality of life outcomes. The goal is to include all pediatric patients undergoing proton therapy and photon therapy to enable future comparisons of treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with either proton or photon radiation therapy.

Exclusion Criteria:

* Greater than 26 years old

Ages: 0 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric brain tumor and bone and soft tissue sarcoma patients that are being treated with proton or photon radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2040-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Approximately 10 years
  Measured from date of diagnosis until death, obtained from medical record notes
Toxicity due to Radiation Therapy as assessed by number of patients with adverse events | Approximately 10 years
  The number of patients that experience adverse events, obtained from medical record notes

CONTACTS AND LOCATIONS:
Overall Officials: Sahaja Acharya, MD, Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland